CLINICAL TRIAL: NCT05071040
Title: Reduction of Sarcopenia Through a Home-based, App-monitored, Physical Exercise Intervention
Brief Title: Sarcopenia and Physical Activity Intervention: a Randomized-controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Scientific Institute San Raffaele (Other)
Collaborators: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Principal Investigator, Paola Cinque, Principal Investigator, Scientific Institute San Raffaele
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RF-2019-12370198
Record Dates: First submitted 2021-09-24; First posted 2021-10-07 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental): Participants will follow a strength exercise program monitored through the use of a specifically designed smartphone application.
  Interventions: Behavioral: Home-based physical activity
- Control group (No Intervention): Continue their daily routine without exercise prescription.

INTERVENTIONS:
Behavioral: Home-based physical activity — Participants will follow a strength exercise program
  Arms: Exercise group

SUMMARY:
Sarcopenia is a pathophysiological process associated with aging and some metabolic conditions characterized by progressive muscle tissue loss, which may lead to loss of strength and performance and increased risk of falls and fractures, physical disability and premature death. With the present project the investigator aim to assess the effect of a feasible exercise program to improve muscle strength (primary outcome), and muscle volume and performance and other measures potentially associated with sarcopenia (secondary outcomes) in elderly and people living with HIV (PLWH) with sarcopenia. The investigators plan to enroll 98 elderly and 98 PLWH in a multicentric, 48-week, randomized, parallel-group, open label, superiority trial comparing the effect of a home-based and app-monitored strength exercise intervention versus no intervention. The investigators expect that participants who exercise will improve strength and other parameters and that improvement at week 12 and week 48 will be higher than in no-exercise controls.

ELIGIBILITY:
Inclusion Criteria:

* Sedentary
* >60 year-old in the elderly group or >50 year-old for the PLWH group;
* with sarcopenia, as defined by both relative loss of muscle mass by bioimpedentiometry (BIA) and low muscle strength by handgrip

Exclusion Criteria:

* Any disease requiring hospitalization in the 6 weeks before enrollment;
* Medical conditions contraindicating the proposed exercise as established by a sport medicine specialist;
* Current substance or alcohol abuse or use of drugs that may influence balance and coordination;
* Not being able to walk without assistance and to perform the prescribed exercises as by protocol.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-10-15 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
Muscle strenght improvement | Week 12
  To assess the effect of exercise on muscle strength assess by the handgrip, in elderly people and PLWH, through comparison between an experimental and a control group.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Ospedale San Raffaele Turro, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided